CLINICAL TRIAL: NCT07102732
Title: VALIDITY AND RELIABILITY OF THE TURKISH VERSION OF THE MODIFIED NEW MOBILITY SCORE
Brief Title: Modified New Mobility Score - Turkish Version
Status: Completed | Type: Observational
Sponsor: Istanbul Rumeli University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other); Fatih Sultan Mehmet Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Ilayda Kayapinar, Research Assistant, Istanbul Rumeli University
Other Study IDs: 2024/10
Record Dates: First submitted 2025-07-30; First posted 2025-08-05 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Hip Fracture; Hip Fracture Surgeries
Keywords: Hip; Fracture; Ambulation; Outcome Measures; Assessment
MeSH Terms: conditions — Hip Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this validation and reliability study is to translate the modified version of the New Mobility Score (NMS) into Turkish (NMS-TR), culturally adapt it, and examine its psychometric properties in elderly individuals (aged 65 years and older) with hip fractures.

The main questions it aims to answer are:

1. Is the New Mobility Score a valid and reliable measurement tool for assessing mobility in Turkish individuals with hip fractures?
2. Is the New Mobility Score not a valid and reliable measurement tool in this population?

There is no comparison group in this study.

Participants will:

Provide demographic and clinical information. Undergo cognitive assessment using the Mini-Mental State Examination (MMSE). Be evaluated for comorbidity burden using the Charlson Comorbidity Index (CCI). Have their ambulatory function assessed with the Cumulative Ambulation Score (CAS).

ELIGIBILITY:
Inclusion Criteria:

* aged 65 years and older
* postoperative hip fracture who were admitted to the Orthopedics and Traumatology Department of Fatih Sultan Mehmet Training and Research Hospital

Exclusion Criteria:

* under the age of 65
* Without a hip fracture
* Not being a voluntary participant

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Voluntary patients aged 65 years and older with a hip fracture
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-21 (Actual); Primary Completion 2025-07-25 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
modified The New Mobility Score | From enrollment, all measurements were repeated within 2 to 7 days following the initial assessment to evaluate test-retest reliability.
  The NMS requires a self-report on the ability to complete walking tasks in different settings, including indoor walking (e.g., within a house), outdoor walking, and walking during shopping. Each item is scored on a scale from 0 to 3 based on the individual's self-reported ability: a score of 0 indicates the individual was unable to complete the task, a score of 1 indicates the individual required assistance from another person to complete the task, a score of 2 indicates the individual completed the task with the aid of a walking aid, and a score of 3 indicates the individual completed the task independently without any walking assistance.
Cumulative Ambulation Score | From enrollment, all measurements were repeated within 2 to 7 days following the initial assessment to evaluate test-retest reliability.
  The Cumulative Ambulation Score assesses four distinct activities (getting out of bed, sitting, and walking) using a three-point ordinal scale ranging from 0 to 2. A score of 0 indicates that the individual is unable to perform the activity despite human assistance and verbal cues; a score of 1 signifies that the activity can be performed with human assistance and/or verbal prompting from one or more individuals; and a score of 2 denotes the ability to perform the activity safely without human assistance or verbal prompting, although the use of a walking aid is permitted. The total score ranges from 0 to 6.

SECONDARY OUTCOMES:
Mini-Mental State Examination | From enrollment, all measurements were repeated within 2 to 7 days following the initial assessment to evaluate test-retest reliability.
  The total score of this test ranges from 0 to 30, with lower scores indicating more pronounced cognitive impairment. In the literature, a cut-off score of 24 is commonly accepted, with scores of 24 or below suggesting a risk of cognitive impairment.
The Charlson Comorbidity Index | From enrollment, all measurements were repeated within 2 to 7 days following the initial assessment to evaluate test-retest reliability.
  The Charlson Comorbidity Index (CCI) is a common tool used to estimate patients' long-term mortality risk. This index plays an important role in assessing health outcomes by measuring the burden of comorbidities that patients have.

CONTACTS AND LOCATIONS:
Overall Officials: İpek YELDAN, PHD PT, Study Director — İstanbul University-Cerrahpaşa
Locations (1):
- Fatih Sultan Mehmet Eğitim ve Araştırma Hastanesi, Istanbul, Ataşehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because participants did not provide explicit consent for data sharing beyond the current study.

REFERENCES:
- [Result] Kristensen MT, Jakobsen TL, Nielsen JW, Jorgensen LM, Nienhuis RJ, Jonsson LR. Cumulated Ambulation Score to evaluate mobility is feasible in geriatric patients and in patients with hip fracture. Dan Med J. 2012 Jul;59(7):A4464. PMID 22759844
- [Result] Parker MJ, Palmer CR. A new mobility score for predicting mortality after hip fracture. J Bone Joint Surg Br. 1993 Sep;75(5):797-8. doi: 10.1302/0301-620X.75B5.8376443.